CLINICAL TRIAL: NCT00551876
Title: A Randomized, Double-Blind, Parallel, Multicenter Study to Evaluate the Efficacy and Safety of Simvastatin Monotherapy Compared With Simvastatin Plus Ezetimibe (SCH 58235) in Type 2 Diabetic Patients Treated With Thiazolidinediones
Brief Title: Study Evaluating the Efficacy and Safety of Simvastatin Alone Compared With Simvastatin Plus Ezetimibe in Type 2 Diabetic Patients (0653-021)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-021; MK0653-021; 2006_554
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ezetimibe; Duration of Therapy; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653, ezetimibe / Duration of Treatment: 30 Weeks
Drug: Comparator : ezetimibe (+) simvastatin / Duration of Treatment: 30 Weeks

SUMMARY:
The purpose of this study is to determine if the addition of ezetimibe 10 mg daily to ongoing 20 mg simvastatin daily will reduce LDL Cholesterol to a greater extent than increasing the dose of simvastatin to 40 mg daily in Type 2 diabetics treated with Thiazolidinediones (TZD).

ELIGIBILITY:
Inclusion Criteria:

* Men or women age between 30 and 75 with Type 2 diabetes mellitus who are treated with pioglitazone or rosiglitazone
* Additionally, patients must have an LDL-C >100 mg/dL at Visit 1 or prior to initiation of statin therapy

Exclusion Criteria:

* Patients taking sliding scale insulin, selected lipid lowering medications, oral anticoagulants and cyclical sex hormones
* Patients with heart disease, kidney disease, liver disease, uncontrolled high blood pressure, and insulin dependent diabetes

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2001-12; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Percent change in fasting LDL-C from baseline to the average of the Week 6/Week 12 measurements | 6 & 12 Weeks

SECONDARY OUTCOMES:
Well tolerated in patients in Diabetic patients | 30 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Gaudiani LM, Lewin A, Meneghini L, Perevozskaya I, Plotkin D, Mitchel Y, Shah S. Efficacy and safety of ezetimibe co-administered with simvastatin in thiazolidinedione-treated type 2 diabetic patients. Diabetes Obes Metab. 2005 Jan;7(1):88-97. doi: 10.1111/j.1463-1326.2004.00420.x. PMID 15642080